CLINICAL TRIAL: NCT07017673
Title: Phase II Trial of Ivonescimab in Combination With Carboplatin + Docetaxel in Patients With Early Stage Triple Negative Breast Cancer
Brief Title: Phase II Trial of Ivonescimab in Combination With Carboplatin + Docetaxel in Patients With Early-Stage Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Principal Investigator, Yuan Yuan, Sponsor-Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024-09-YUAN-NeoIVO
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: TNBC; TNBC - Triple-Negative Breast Cancer; Early Stage Triple-Negative Breast Carcinoma
Keywords: Ivonescimab; Carboplatin; Docetaxel; Neoadjuvant chemotherapy; TNBC; High-risk early stage TNBC
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carboplatin and Ivonescimab (Experimental): Carboplatin AUC6 and docetaxel 75 mg/m2 every 3 weeks x 6 cycles plus ivonescimab 20 mg/kg iv every 3 weeks x 6 cycles. Each cycle is 21 days. Trial interventions may be administered up to 3 days before or after the scheduled Day 1 of each cycle due to administrative reasons (after all safety assessments have been completed).
  Interventions: Drug: Ivonescimab; Drug: Carboplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Ivonescimab — Drug: Ivonescimab Dose: 20 mg/kg Route: IV infusion over 60 minutes Frequency: Q3W Duration: 6 cycles (Each cycle is 21 days)
Drug: Carboplatin — Drug: Carboplatin Dose: AUC6 Route: IV infusion Frequency: Q3W Duration: 6 cycles (Each cycle is 21 days)
Drug: Docetaxel — Drug: Docetaxel Dose: 75 mg/m^2 Route: IV infusion over 60 minutes Frequency: Q3W Duration: 6 cycles (Each cycle is 21 days)

SUMMARY:
This is a single arm phase II trial combination of ivonescimab and carbo-docetaxel every 3 weeks for 6 cycles in patients with early-stage triple negative breast cancer. The trial is designed to test the safety and efficacy of adding ivonescimab in patients with early TNBC undergoing neoadjuvant chemotherapy with carboplatin and docetaxel. Patients will receive ivonescimab 20 mg/kg IV on Day 1 of each cycle, and carboplatin AUC6 and docetaxel 75 mg/m2 on Day 1 of each cycle for 6 cycles. Cycles will be 21 days for a total of 6 cycles. Curative intent surgery will be performed within 6 weeks (maximum 12 weeks) time frame upon completion of last dose of chemoimmunotherapy. The surgical pathology information will be used for assessment of pathological response, which serve as the primary endpoint of this study. Patients will undergo assessment at baseline, C1D1 of each cycle and end of treatment visit for collection of treatment-emergent adverse events, evaluated by CTCAE v5.0. Patient reported outcomes will be collected at cycles 1, 4, and 6, and at EOT. All study patients will be followed for at least 5 years for EFS and OS follow up. Research biopsies, peripheral blood and stool samples will be collected at the following time points: baseline, C4D1 (+/-14 days), and surgery (+/-14 days). Baseline and EOT breast MRI will be performed as standard of care for assessment of clinical response. Mid treatment breast ultrasound (C4D1 +/-14 days) will be repeated as standard of care to assess clinical response to treatment. Mid-treatment C4D1 tumor biopsy may be omitted if the primary tumor is no longer visible or the tumor deemed too small for biopsy by radiologist.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years of age
* ECOG ≤ 1
* High-risk early stage triple negative breast cancer (TNBC), defined by ER≤10%, PR≤10% and HER2 negative (by IHC or FISH), per ASCO/CAP guidelines
* Clinically ≥T1cN0, or any T, N1-2
* Plan to receive neoadjuvant chemotherapy and immune checkpoint inhibitor before surgery as standard-of-care treatment
* Adequate organ function as defined in the following. Specimens must be collected within 14 days prior to the start of study treatment.

  * ANC ≥ 1,500/mm3
  * Platelets ≥ 100,000/mm3
  * Hemoglobin ≥ 9.0 g/dL.
  * Total serum bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 x ULN
  * AST < 3 x ULN
  * ALT < 3 x ULN
  * Creatinine clearance ≥ 30 mL/min
  * INR or PT, aPTT < 1.5 x ULN
* Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test within 14 days of start of study treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: If egg harvesting was completed prior to enrollment, the pregnancy test may be falsely positive and the PI will assess and determine eligibility for these cases.
* Female participants: A female participant is eligible to participate if she is not pregnant (see Appendix B), not breastfeeding, and at least one of the following conditions applies:

  -- Not a woman of childbearing potential (WOCBP) as defined in Appendix B OR Females of child-bearing potential must be willing to use effective contraception during study and for 120 days after the last dose.
* Male participants: A male participant must agree to use a contraception as detailed in Appendix B of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria

* Evidence of metastatic disease.
* Is currently participating in or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to start of study treatment, including but not limited to:

  * Hemoptysis (defined as coughing up ≥ 0.5 teaspoon of fresh blood or small blood clots) Note: transient hemoptysis associated with diagnostic bronchoscopy is allowed.
  * Nasal bleeding/epistaxis (bloody nasal discharge is allowed)
  * Current use of prophylactic or full-dose anticoagulants or anti-platelet agents for therapeutic purposes that is not stable, in the opinion of the treating investigator, prior to start of study treatment is not allowed. The use of full-dose anticoagulants is permitted as long as the INR or activated partial thromboplastin time (aPTT) is within therapeutic limits according to the medical standard of the enrolling institution.
* Poorly controlled hypertension with repeated systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg after oral antihypertensive therapy
* Women who are or are planning to become pregnant or breastfeed
* Known allergy to any of the components within the study agents and/or their excipients
* Medical history and concurrent diseases

  * Autoimmune diseases
  * Any prior malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for at least three years
  * History of (non-infectious) pneumonitis that required steroids or has current pneumonitis
  * Active infection requiring systemic therapy
  * Known history of Human Immunodeficiency Virus (HIV) infection
  * Known history of active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority
  * Known history of active TB (Mycobacterium tuberculosis)
  * History of unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] classification ≥ grade 2) or unstable vascular disease (eg, aortic aneurysm at risk of rupture, Moyamoya disease) that required hospitalization within 12 months prior to randomization, or other cardiac impairment that may affect the safety evaluation of the study drug (eg, poorly controlled arrhythmias, myocardial ischemia)
  * Prolongation of QTc interval >480 msec
  * Prior allogeneic bone marrow transplantation or prior solid organ transplantation
  * History of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months prior to start of study treatment
  * History of any grade arterial thromboembolic event, Grade 3 and above venous thromboembolic event, as specified in National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 12 months prior to start of study treatment
  * Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks before start of study treatment
  * History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to start of study treatment
* Prohibited Treatments and/or Therapies

  * Other non-protocol specified anti-cancer therapy: systemic radiotherapy, immunotherapy, biologic, or hormonal therapy. tretinoin therapy, nitrosourea, mitomycin C, small molecule tyrosine kinase inhibitor therapy

    --- Concomitant use of hormones for non-tumor-related conditions (e.g., insulin and hormone replacement therapy for diabetes mellitus) is acceptable
  * Any live vaccine within 30 days prior to the first dose of study drug and up to 120 days after the last dose. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed
  * Prior systemic therapy or radiation therapy with curative intent for the current breast cancer
  * A previous definitive ipsilateral breast surgery for the current breast cancer
  * Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. CTLA-4, OX-40, CD137).
  * Immunosuppressive drugs, including, but not limited to, prednisone or equivalent, methotrexate, azathioprine, and TNF-α antagonists at doses exceeding 10 mg per day. The following exceptions are allowed:

    * The use of immunosuppressive drugs for the treatment of study drug-associated AEs or the use of immunosuppressive drugs in subjects with contrast allergy is acceptable.
    * The use of inhaled, topical, and intranasal glucocorticoids is permitted.
    * Corticosteroids are allowed as a prophylactic drug for hypersensitivity reactions (eg, before CT or MRI).
    * Corticosteroids are allowed as antiphylactic and therapeutic agents for chemotherapy-induced vomiting.
    * Short-term use of glucocorticoids for underlying or intercurrent conditions may be permitted after discussion with the PI.
* Major surgery within 28 days prior to start of study treatment and within 4 weeks after first dose. Participants must have fully recovered from the effects of prior major surgery in the opinion of the treating investigator.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | 6 months (From cycle 1 day 1 till surgery)
  Pathological complete response (pCR) will be defined as the absence of invasive disease in the breast and lymph nodes at the time of SOC curative-intent surgery. This will be assessed at time of surgery. Pathological responses will be evaluated using residual cancer burden (RCB) classifier defined by ASCO/CAP guideline.

SECONDARY OUTCOMES:
To determine the overall safety of ivonescimab in combination with carboplatin and docetaxel in patients with early-stage TNBC by CTCAE v5.0. | 9 months (From Cycle 1 until 90 days post last dose of study treatment)
  Frequency and severity of treatment-emergent adverse events, evaluated by CTCAE v5.0.
Event-free survival (EFS) | From cycle 1 day 1 till end of follow up (up to 5 years)
  Event-free survival (EFS) measured from start of study treatment to the first occurrence of recurrent disease, or death due to breast cancer.
Overall survival (OS) | From cycle 1 day 1 till end of follow up (up to 5 years)
  Overall survival (OS) measured from start of study treatment to death or last contact (censored)
Patient-reported outcomes (PRO) | 9 months
  Patient-reported outcomes (PRO) will be measured by changes in the PROMIS-29 Profile physical function subscale score measured at start of study treatment and End of Treatment.
  The PROMIS-29 scoring provides T-scores that indicate the level of a patient's health-related quality of life compared to a reference population. A T-score of 50 represents the average score for that population. Higher scores generally indicate more of the concept being measured, such as physical function or mental health.
Patient-reported outcomes (PRO) | 9 months
  Patient-reported outcomes (PRO) will be measured by changes in the PROMIS Fatigue 7a measured at start of study treatment and End of Treatment. The PROMIS 7a scoring system uses a standardized T-score with a mean of 50 and a standard deviation of 10, allowing for comparison of individuals to the general population. A higher T-score generally indicates a higher level of the specific trait being measured (e.g., fatigue, anxiety, depression).

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Yuan, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (4):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center Beverly Hills, Los Angeles, California
  - Huntington Cancer Center, an Affiliate of CS Cancer, Pasadena, California
  - Hunt Cancer Institute, an Affiliate of CS Cancer, Torrance, California